CLINICAL TRIAL: NCT00825864
Title: Evaluation the Effect of Diclofenac Drops vs Dexamethasone Drops in Trabeculectomy and Cataract Surgery
Brief Title: Diclofenac vs Dexamethasone in Combined Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Levkovitch-Verbin Hani, Goldschleger Eye Institute, Sheba Medcial Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-03-3123-HLV-CTIL
Record Dates: First submitted 2009-01-18; First posted 2009-01-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Glaucoma; Cataract
MeSH Terms: conditions — Glaucoma; Cataract | interventions — dexamethasone 21-phosphate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1diclofenac drops treatment (Active Comparator): four times a day for 3 months
  Interventions: Drug: diclofenac drops
- 2dexamethasone drops (Active Comparator)
  Interventions: Drug: dexamethasone sodium phosphate 0.1% eye drops

INTERVENTIONS:
Drug: diclofenac drops — one drop 4 times a day for 3 months
  Arms: 1diclofenac drops treatment
Drug: dexamethasone sodium phosphate 0.1% eye drops — for first week after the operation : one drop 6 times a day. Then tapering by reducing one drop for a week
  Arms: 2dexamethasone drops

SUMMARY:
To study the effect of Diclofenac drops or Dexamethasone drops on combined surgery of trabeculectomy and cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for combines surgery of trabeculectomy and cataract surgery

Exclusion Criteria:

* severe complicated surgery like vitreal loss, expulsive hemorrhage, endophthalmitis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | year

SECONDARY OUTCOMES:
the number of antiglaucoma medications | year

CONTACTS AND LOCATIONS:
Overall Officials: Hani Levkovitch-Verbin, Principal Investigator — Tel-Aviv University, Israel
Locations (1):
- Goldschleger Eye Institute, Sheba Medcial Center, Tel Litwinsky, Israel